CLINICAL TRIAL: NCT02100735
Title: Evaluation of an Analgosedation Protocol in Mechanically Ventilated Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in with enrollment of patient
Sponsor: Tampa General Hospital (Other)
Responsible Party: Principal Investigator, Beatrice Adams, Pharmacotherapy Specialist, Tampa General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00016830
Record Dates: First submitted 2014-03-21; First posted 2014-04-01 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Effect of Protocolized Sedation on Days of Mechanical Ventilation in the ICU
Keywords: sedatives; analgesics; protocol; mechanical ventilation; analgosedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation protocol (Experimental): Sedation protocol is a document that will be used to guide the adjustment of sedation in the ICU.
  Interventions: Other: Sedation protocol
- Standard of care (Active Comparator): Current practices
  Interventions: Other: Sedation protocol

INTERVENTIONS:
Other: Sedation protocol — Nursing driven sedation protocol
  Other Names: The sedation protocol is a document that wil lbe used by healthcare providers to guide sedation used in the ICU

SUMMARY:
The purpose of this study is to evaluate how the investigators provide sedation (medicine that make you sleepy) in the investigators intensive care unit (ICU). This study will look at a new way of using sedation in the ICU to see what effect it has on patients and if it decreases the amount of time spent on mechanical ventilation (machine that breathes for you), and in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients expected to require mechanical ventilation for greater than 48 hrs

Exclusion Criteria:

* Need for continuous neuromuscular blockade
* Severe chronic neurocognitive dysfunction
* Tracheostomy at the time of study enrollment
* Alcohol withdrawal risk or symptoms
* Drug overdose
* Chronic use of narcotics
* Active seizures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Days on mechanical ventilation | Participants will be assessed daily for the duration of their stay in the ICU, an expected average of 4-5 days

SECONDARY OUTCOMES:
ICU Length of stay | Participants will be followed for the entire length of their ICU stay, expected average of 4-7 days
28 day mortality | Participants will be followed for 28 days from enrollment into the study

CONTACTS AND LOCATIONS:
Locations (1):
- Beatrice Adams, Riverview, Florida, United States